CLINICAL TRIAL: NCT05461365
Title: Intranasal Insulin for COVID-19-related Smell Loss
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad Panamericana (Other)
Responsible Party: Principal Investigator, Daniel Dibildox Reynoso, Professor, Universidad Panamericana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01007
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Anosmia; Smell Loss; Paraosmia; Hyposmia; COVID-19
MeSH Terms: conditions — Anosmia; Olfaction Disorders; COVID-19 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intranasal insulin (Experimental): For each selected participant (n=27), a baseline olfactory measurement was performed with Sniffin Sticks® (12 items) and a capillary glucose measurement was obtained with Dextrostix® NF before and after the intervention, in order to guarantee patient safety and reduce the risk of hypoglycemia. The initial and final measurements were divided into three subsections with a different number of correct answers for each section Subsequently, Gelfoam® cottonoids soaked in 40 IU of NPH insulin were placed on the nasal roof (between the nasal septum and the middle meatus) of each nostril. These remained in place for 15 minutes and were later removed. This procedure was performed in three visits one week apart. During the fourth and last visit (one week after the previous visit), olfaction was reevaluated using the measures previously described.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Gelfoam® cottonoids soaked in 40 IU of NPH insulin were placed on the nasal roof (between the nasal septum and the middle meatus) of each nostril. These remained in place for 15 minutes and were later removed. This procedure was performed in three visits one week apart. During the fourth and last visit (one week after the previous visit), olfaction was reevaluated using the measures previously described.
  Other Names: intranasal insulin

SUMMARY:
The aim of this study was to quantify the improvement in olfaction of 27 post-COVID-19 patients, after three intreventions of intranasal insulin during a four week period, with the help of the Threshold, Discrimination and Identification (TDI) score evaluated with Sniffin Sticks®.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 in the last 3 to 18 months and who persisted with anosmia, hyposmia or other olfactory dysfunction chronically and without improvement

Exclusion Criteria:

* nasal tumors, chronic sinusitis, drug-induced sinusitis, nasal polyposis, neurodegenerative disease, smoking, pregnancy Hypoglycemia and a previous diagnosis of diabetes mellitus or anatomical malformations such as septal deviation, rhinosinusitis or choanal atresia

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
SMELL LOSS IMPROVEMENT | 1 MONTH

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Panamerican, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Oleszkiewicz A, Schriever VA, Croy I, Hahner A, Hummel T. Updated Sniffin' Sticks normative data based on an extended sample of 9139 subjects. Eur Arch Otorhinolaryngol. 2019 Mar;276(3):719-728. doi: 10.1007/s00405-018-5248-1. Epub 2018 Dec 15. PMID 30554358
- [Background] Kosugi EM, Lavinsky J, Romano FR, Fornazieri MA, Luz-Matsumoto GR, Lessa MM, Piltcher OB, Sant'Anna GD. Incomplete and late recovery of sudden olfactory dysfunction in COVID-19. Braz J Otorhinolaryngol. 2020 Jul-Aug;86(4):490-496. doi: 10.1016/j.bjorl.2020.05.001. Epub 2020 May 25. PMID 32534982
- [Background] Vaira LA, Salzano G, Fois AG, Piombino P, De Riu G. Potential pathogenesis of ageusia and anosmia in COVID-19 patients. Int Forum Allergy Rhinol. 2020 Sep;10(9):1103-1104. doi: 10.1002/alr.22593. Epub 2020 Jun 15. No abstract available. PMID 32342636
- [Result] Rezaeian A. Effect of Intranasal Insulin on Olfactory Recovery in Patients with Hyposmia: A Randomized Clinical Trial. Otolaryngol Head Neck Surg. 2018 Jun;158(6):1134-1139. doi: 10.1177/0194599818764624. Epub 2018 Mar 20. PMID 29557250
- [Result] Mohamad SA, Badawi AM, Mansour HF. Insulin fast-dissolving film for intranasal delivery via olfactory region, a promising approach for the treatment of anosmia in COVID-19 patients: Design, in-vitro characterization and clinical evaluation. Int J Pharm. 2021 May 15;601:120600. doi: 10.1016/j.ijpharm.2021.120600. Epub 2021 Apr 14. PMID 33862126